CLINICAL TRIAL: NCT00169520
Title: A Phase I, Open-Label Study of SB-715992 in Combination With Docetaxel in Patients With Advanced Solid Tumors.
Brief Title: SB-715992 In Combination With Docetaxel In Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSP10003
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Solid Tumor Cancer
Keywords: Safety; tolerability; dose limiting toxicity; solid tumors; docetaxel
MeSH Terms: interventions — Docetaxel; ispinesib

INTERVENTIONS:
Drug: docetaxel
Drug: SB-715992
  Other Names: docetaxel

SUMMARY:
The purpose of this study is to determine the dose regimen of SB-715992 in combination with docetaxel in patients with solid tumors. SB-715992 and docetaxel were dosed by 1-hour intravenous infusion every 3 weeks (on the same day). A patient may continue to receive treatment as long as they are benefiting from the treatment. Blood samples will be taken at specific times to measure the amount of both drugs in your body at specific times after the drug is given. Blood samples will also be taken for lab tests such as complete blood counts and clinical chemistries. Physical exams will be performed before each treatment with SB-715992. During the treatment phase, the patients will undergo regular assessments for safety and clinical response.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of an advanced solid tumor malignancy that is not responsive to standard therapies or for which there is no standard therapy.
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0-2.

Exclusion criteria:

* Females who are pregnant or nursing.
* Pre-existing hemolytic anemia.
* Pre-existing peripheral neuropathy greater than or equal grade 2. Greater than or equal to 4 prior chemotherapy regimens including neoadjuvant/adjuvant chemotherapy, except breast cancer subjects who may have received more than 4 prior chemotherapy regimens.
* Absolute neutrophil count less than 1,500/mm3.
* Platelets less than 100,000/mm3.
* Hemoglobin less than 9 g/dL.
* Total bilirubin greater than1.5 mg/dL.
* AST/ALT greater than 2.5 X upper limit of normal.
* Creatinine clearance less than or equal to 60 mL/min (calculated by the Cockcroft Gault Formula).
* Known contraindications to the use of docetaxel or to other drugs formulated with polysorbate 80.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-06

PRIMARY OUTCOMES:
Safety and tolerability endpoints will consist of the valuation of adverse events (AEs),vital signs and laboratory values. A dose regimen where 1 of 6 (or 17%) subjects experience a dose-limiting toxicity. | throughout the study

SECONDARY OUTCOMES:
PK endpoints of SB-715992 and docetaxel pending the conduct of the PK interaction portion. Antitumor activity will be assessed every 2 cycles (PD). | every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Oxford, Oxfordshire
  - GSK Investigational Site, London